CLINICAL TRIAL: NCT05622916
Title: The Efficacy of Ethanol Extract of Red Betel Leaves (Piper Crocatum) as Topical Patient-Applied Therapy In Anogenital Warts The Study of Foxp3+ Treg, Tumor Growth Factor (TGF)-β1, and Interferon (IFN)-γ Expression
Brief Title: Topical Ethanol Extract (Piper Crocatum) for Anogenital Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1114222112
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Anogenital Wart
Keywords: Anogenital Wart; Trichloroacetic; Piper crocatum; Clinical Efficacy; Inflammatory Marker
MeSH Terms: conditions — Condylomata Acuminata | interventions — Ethanol; Trichloroacetic Acid

STUDY DESIGN:
Intervention Model Description: One group will receive the intervention, whereas the comparison group will receive standard care
Who Masked: Participant
Masking Description: participants will be blind from the allocation by mimicking the topical solution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Daily topical application (twice/day, in the morning and 30-60 minutes before bed at night) for 56 days.
  Interventions: Drug: Topical Ethanol Extract (Piper crocatum)
- Comparison (Active Comparator): Weekly application (1x/week) by the physician for 8 weeks
  Interventions: Drug: Trichloroacetic Acid Topical

INTERVENTIONS:
Drug: Topical Ethanol Extract (Piper crocatum) — Topical ethanol extract of red betel leaves (Piper crocatum) 30% with the details of formulation on detailed description section
  Other Names: Red Betel Leaves
  Arms: Intervention
Drug: Trichloroacetic Acid Topical — Trichloroacetic acid topical 90%
  Other Names: TCA 90
  Arms: Comparison

SUMMARY:
This clinical trial aims to assess the efficacy of topical Piper crocatum in treating Anogenital warts. It aims to answer

* the clinical efficacy of treating anogenital warts
* the expression of Foxp3+ regulatory T (Treg), TGF/Tumor Growth Factor -β1, and IFN/interferon -γ of anogenital wart lesion Participants will be allocated into two topical treatments, intervention and active comparator Trichloroacetic Acid (TCA) 90%. The researchers assume that intervention is superior compared to TCA 90%

DETAILED DESCRIPTION:
Study Design :

A randomized controlled trial

Population:

Diagnosed with Condyloma Acuminata (International Classification of Disease 10 code A.63.0)

Intervention period :

8 weeks of daily topical intervention with follow-up at week 12

Detailed formulation

1. Extraction of Piper crocatum with ethanol assisted in a microwave-assisted extraction (MAE)
2. The dissolution and active substances are separated by evaporation using a rotary evaporator to obtain the extract in the form of a thick solution
3. freeze-drying is performed to obtain a stable thick extract
4. preparation of ointment by adding formulation of ethanol extract of red betel leaves with 50 mg of white vaseline to achieve 30% concentration

Settings:

Outpatient care at the designated hospital

Participants:

Consecutive recruitment

Sample Size Estimation:

Following the formula of two different means, with the indicator, as follows:

1. Type 1 error 5%
2. Power of Study 80%
3. Assuming the effect size of cohen d (in reducing the size of warts) is 0.5
4. equal allocation between two arms total sample: 100 participants

Proposed analysis:

Intention to treat (ITT) with sensitivity and subgroup analysis

ELIGIBILITY:
Inclusion Criteria:

1. Men and women diagnosed with external anogenital warts
2. Clinical lesions of Anogenital Wart at least 3 lesions with a size of 1-5 cm
3. In patients with HIV, Cluster of Differentiation 4 (CD4)cell count >350 cells/mm and have been taking antiretroviral (ARV) drugs regularly for 3 months,

Exclusion Criteria:

1. Pregnant or lactating women
2. Lesions located in the external urethral orifice and vagina
3. Using systemic immunomodulators/immunosuppressants

The protocol treatment will be discontinued if patients

a. Withdraw their consent based on the patient's demand d. Severe adverse events occurred or allergies to the components of the test product b. After undergoing clinical trials, the patient experienced things that caused him/her to no longer meet the criteria set out in this protocol. c. Subjects do not comply the established study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Size of wart | Changes of wart size from baseline to week 12
  the size of wart measured from the outermost edge of the warts.
Foxp3+ regulatory T (Treg) | change of Foxp3+ regulatory T (Treg) expression from baseline to week 8
  the expression of Foxp3+ regulatory T (Treg) from the stained T cells in anogenital wart lesion
TGF-β1 | change of TGF-β1 expression from baseline to week 8
  the expression of TGF-β1 from the stained cells in anogenital wart lesion
IFN-γ | change of IFN-γ expression from baseline to week 8
  the expression of IFN-γ from the stained cells in anogenital wart lesion

OTHER OUTCOMES:
Adverse reaction | any adverse event from baseline to week 12
  any records of adverse reaction including inflammation, irritation or other systemic adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Idrianti Idrus, MD, Principal Investigator — Hasanuddin University; Wresti Indriatmi, MD. Ph.D, Principal Investigator — Indonesia University; Fransiscus Suyatna, MD. Ph.D, Principal Investigator — Indonesia University
Locations (1):
- Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
de-identified data will be shared for specific purpose, including article review

REFERENCES:
- [Background] Sherrard J, Riddell L. Comparison of the effectiveness of commonly used clinic-based treatments for external genital warts. Int J STD AIDS. 2007 Jun;18(6):365-8. doi: 10.1258/095646207781024711. PMID 17609022
- [Background] Gilson R, Nugent D, Werner RN, Ballesteros J, Ross J. 2019 IUSTI-Europe guideline for the management of anogenital warts. J Eur Acad Dermatol Venereol. 2020 Aug;34(8):1644-1653. doi: 10.1111/jdv.16522. PMID 32735077
- [Background] Sazwi NN, Nalina T, Abdul Rahim ZH. Antioxidant and cytoprotective activities of Piper betle, Areca catechu, Uncaria gambir and betel quid with and without calcium hydroxide. BMC Complement Altern Med. 2013 Dec 11;13:351. doi: 10.1186/1472-6882-13-351. PMID 24330738
- [Background] Pharm T, Hartini YS, Wahyuono S, Widyarini S, Yuswanto A. Hartini et al In vivo Immunomodulatory Effect and Histopathological Features of Mouse Liver and Kidney Treated with Neolignans Isolated from Red Betel (Piper crocatum Ruiz & Pav) Leaf. Tropical Journal of Pharmaceutical Research. 2014;13:1609-1614. doi:10.4314/tjpr.v13i10.6
- [Background] Bonin CM, Padovani CTJ, da Costa IP, Avila LS, Ferreira AMT, Fernandes CES, Dos Santos AR, Tozetti IA. Detection of regulatory T cell phenotypic markers and cytokines in patients with human papillomavirus infection. J Med Virol. 2019 Feb;91(2):317-325. doi: 10.1002/jmv.25312. Epub 2018 Sep 24. PMID 30192406
- [Background] Xu Y, Zhu KJ, Zhu N, Jiang DH, Chen XZ, Cheng H. Expression of Foxp3+CD4+CD25+ regulatory T cells and Th1/Th2, Tc1/Tc2 profiles in the peripheral blood of patients with condyloma acuminatum. Clin Exp Dermatol. 2009 Mar;34(2):229-35. doi: 10.1111/j.1365-2230.2008.03001.x. Epub 2008 Dec 2. PMID 19077104